CLINICAL TRIAL: NCT01679444
Title: Magnetic Resonance Spectroscopy Probe Study of Alcohol Use
Brief Title: MRS Probe Study of Alcohol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Frye, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 12-003693
Record Dates: First submitted 2012-08-30; First posted 2012-09-06 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Heavy Dose Drinkers
Keywords: MRS; Heavy dose drinkers; Alcohol; NIAAA
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopy
  Other Names: MRS

SUMMARY:
This protocol will investigate the neurobiological underpinnings of alcohol craving in recently detoxified alcoholic drinkers utilizing novel functional brain imaging. This clinical magnetic resonance spectroscopy (MRS) study will investigate whether glutamate and other brain metabolites correlate to measures of alcohol craving severity

ELIGIBILITY:
Inclusion Criteria: (Minimal or No Alcohol Group)

1. Male or female age 21-70
2. Consume less alcohol then what is described in this protocol as a "higher dose drinker", or consume no alcohol at all.
3. Able to complete a 60 min. MRS brain scan.

Exclusion Criteria:

1. Inability to speak English
2. Inability or unwillingness to provide written informed consent
3. Diagnosis of active substance dependence other than nicotine (e.g. alcohol, cannabis, caffeine, prescription use of barbiturates, benzodiazepines, opiates, or stimulants) this will be determined using a PRISM (Psychiatric Research Interview for Substance and Mental Disorders) interview.
4. Any unstable active medical or additional psychiatric condition as determined by the investigator
5. Active suicidal ideation as determined by the PHQ-9 question 9 indicating response #2 or higher (several days; more than half the days; or nearly every day).
6. History of encephalopathy, hepatic failure, or HIV seropositivity
7. History of claustrophobia
8. History of major head trauma with loss of consciousness >5 minutes or skull fracture
9. History of previous neurological event (e.g. epilepsy, stroke, transient ischemic attack)
10. Implanted metal objects (e.g. pacemakers; aneurysm clips; metal prostheses, joints, rods, or plates)
11. Contraindication to MRI scanning
12. Pregnancy or breast-feeding

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Utilizing Magnetic Resonance Spectroscopy at 3 Tesla, investigate the neurobiological underpinnings of alcohol craving
  assessing baseline perturbations in anterior cingulate and ventral striatal metabolites (NAA levels, glutamate levels, glutamine levels)

SECONDARY OUTCOMES:
Evaluate the relationship between these metabolites, each reported as a Cerebrospinal Fluid-corrected absolute concentration, and severity of alcohol cravings
  Evaluate the relationship between these metabolites, each reported as a Cerebrospinal fluid-corrected absolute concentration, and severity of alcohol cravings, as measured primarily by the Penn Alcohol Craving Scale and secondarily by the Inventory of Drug Taking Situations.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States